CLINICAL TRIAL: NCT00225069
Title: Thoracoscopic Sympathectomy for Blushing. A Prospective Randomised Trial.
Brief Title: Thoracoscopic Sympathectomy for Blushing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Peter B Licht, Professor, Odense University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TOPSY1-2005
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Facial Blushing
Keywords: Facial blushing; Sympathectomy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): T2 sympathectomy
  Interventions: Procedure: Level of sympathectomy
- 2 (Experimental): T2-T3 sympathectomy
  Interventions: Procedure: Level of sympathectomy

INTERVENTIONS:
Procedure: Level of sympathectomy — T2 sympathectomy or T2-T3 sympathectomy

SUMMARY:
To determine outcome and side effects following thoracoscopic sympathectomy in patients treated for disabling isolated facial blushing and investigate if there are any significant differences between two different routine procedures: T2 or T2-T3 sympathectomy.

DETAILED DESCRIPTION:
To determine the outcome and side effects following thoracoscopic sympathectomy in patients treated for disabling isolated facial blushing. In addition, following randomization investigate if there are any significant differences between two different routine procedures: T2 or T2-T3 sympathectomy. Includes QoL before and 12 months after surgery

ELIGIBILITY:
Inclusion Criteria:

* Isolated disabling facial blushing
* Over 18 years of age
* Willing to be randomized

Exclusion Criteria:

* Primary hyperhidrosis in palms or axillae
* Previous lung surgery
* Bradycardia
* Arrythmias
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Effect of operation. Side effects: compensatory and gustatory sweating. | 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Licht, MD PhD, Principal Investigator — Odense University Hospital; Hans K Pilegaard, MD, Study Chair — Skejby Sygehus, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Dept Cardiothoracic Surgery, Skejby Sygehus, Aarhus University Hospital, Aarhus
  - Dept Cardiothorcic Surgery, Odense University Hospital, Odense